CLINICAL TRIAL: NCT02326285
Title: Induction Therapy With Gefitinib Followed by Taxane Platinum Chemotherapy and Intercalated Gefitinib in NSCLC Stages II-IIIB With Activating EGFR Mutation - A Single Arm Phase II Trial.
Brief Title: Induction Therapy With Intercalated Tyrosine Kinase Inhibitor (TKI) and Chemotherapy in NSCLC With Activating Epidermal Growth Factor Receptor (EGFR) Mutation in Stages II-IIIB
Acronym: NeoIntercal
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to low patient enrollment was stopped. Only one patient could be enrolled. 37 patients were pre-screened, but not into the inclusion criteria (wt-EGFR)
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-TRK-0214; 2014-005595-28 (EudraCT Number); IISR ESR-14-10598 (Other: AstraZeneca)
Record Dates: First submitted 2014-12-18; First posted 2014-12-29 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Non-squamous Non-small Cell Lung Cancer Stage II; Non-squamous Non-small Cell Lung Cancer Stage IIIA; Non-squamous Non-small Cell Lung Cancer Stage IIIB; Activating EGFR Mutation; NSCLC
Keywords: induction therapy; NSCLC; Non-small Cell Lung Cancer; curative surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Docetaxel; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment phase (Experimental): Enrolled patients will be treated with 250mg/day Gefitinib for 11 days (day -12 until day -1) followed by 3 cycles (length 21 days) of chemotherapy with docetaxel (75mg/m2 d1) and cisplatin (50 mg/m2 d1+2) combined with intercalated gefitinib (250mg/day, d4-20 (cycle 1 and 2) and d4-17 (for cycle3). Surgery is planned in the 4th week after d1 of the last cycle.
  Interventions: Drug: Gefitinib; Drug: docetaxel; Drug: cisplatin; Procedure: Surgery

INTERVENTIONS:
Drug: Gefitinib — Patients will be treated for 12 days with gefitinib 250 mg/day p.o. (d -12 to -1) and induced with chemotherapy docetaxel 75 mg/m2 and cisplatin 50 mg/m2 d1+2 and intercalated gefitinib 250 mg/day d4-20 (cycle 1 and 2) and d4-17 (for cycle3). Surgery is planned in the 4th week after d1 of the last cycle.
  Other Names: IRESSA ®
Drug: docetaxel — chemotherapy docetaxel 75 mg/m2 and cisplatin 50 mg/m2 d1+2 and intercalated gefitinib 250 mg/day d4-20 (cycle 1 and 2) and d4-17 (for cycle3).
Drug: cisplatin — chemotherapy docetaxel 75 mg/m2 and cisplatin 50 mg/m2 d1+2 and intercalated gefitinib 250 mg/day d4-20 (cycle 1 and 2) and d4-17 (for cycle3).
Procedure: Surgery — Surgery should be performed in the 4th or at the latest 5th week after d1 of the last cycle of chemotherapy (d64 to 78).

SUMMARY:
This study is designed as a single arm, un-controlled, open-label, multi-center hypothesis generating two-stage phase II trial. It is based on the assumption that the proposed treatment scheme doubles the rate of pathologic complete remission in Mutated epidermal growth factor receptor (EGFRmt) + NSCLC patients compared to historical control data from standard treatments.

Patients with NSCLC and activating EGFR mutation in stages II, IIIA and IIIB eligible for induction therapy with docetaxel and cisplatin and gefitinib

Patients will be treated for 12 days with gefitinib 250 mg/day p.o. (d -12 to -1) and induced with chemotherapy docetaxel 75 mg/m2 and cisplatin 50 mg/m2 d1+2 and intercalated gefitinib 250 mg/day d4-20 (cycle 1 and 2) and d4-17 (for cycle3). Surgery is planned in the 4th week after d1 of the last cycle.

DETAILED DESCRIPTION:
Based on the notion that neoadjuvant combination of Chemotherapy (CTx) and intercalated TKI is clinically beneficial, which can be inferred from prior study data and single case reports, this study aims to generate additional information on feasibility, safety and efficacy of this treatment approach in a larger group of EGFR mutated NSCLC patients. This study is a hypothesis generating two-stage trial for future phase III studies of neoadjuvant CTx with intercalated TKI. Hence, the study design relies entirely on a single treatment arm. To demonstrate efficacy it is sufficient to compare to historical data of the conventional treatments of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed non-squamous non-small-cell lung cancer (NSCLC) stage II, IIIA and IIIB detected preoperatively by adequate methods and activating EGFR mutation in exons 18-21 and deemed to be able to undergo curative surgery after induction therapy. Stage should be confirmed by PET-CT as well as adequate mediastinal staging. MRI of the brain to exclude CNS metastases is mandatory.
2. At least one unidimensionally measurable lesion meeting RECIST criteria (version 1.1);
3. Performance status of 0 to 1 on the ECOG scale;
4. Estimated life expectancy of at least 12 weeks;
5. Patients aged ≥ 18 years;
6. Adequate organ function including the following:

   1. Adequate bone marrow reserve:

      * absolute neutrophils (segmented and bands) count (ANC) ≥1.5x109/L;
      * platelets ≥100x109/L;
      * haemoglobin ≥9 g/dL.
   2. Hepatic:

      * bilirubin ≤ 1xULN;
      * alkaline phosphatase (AP);
      * aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5xULN.
   3. Renal:

      * serum creatinine ≤ 1.3 mg/dL
      * glomerular filtration rate (GFR) ≥ 70 mL/min for cisplatinum based CTx;
      * If contraindications including GFR below 70mL/minagainst cisplatin exist, carboplatin may also be used;
      * glomerular filtration rate ≥ 30 mL/min (calculated) if carboplatin is to be used
7. Adequate lung function tests as assessed by body plethysmography, diffusion test and if necessary spiro-ergometry.
8. Cooperation and willingness to complete all aspects of the study;

   * Written informed consent to participate in the study.

Exclusion Criteria:

1. EGFR wild type configuration;
2. EGFR resistance mutations (i.e. T790M);
3. Significant cardiovascular disease, such as uncontrolled hypertension, myocardial infarction within the last 6 months, unstable angina pectoris, CHF ≥ NYHA 2, serious arrhythmia, significant peripheral vascular disease;
4. Pre-existing neuropathic ≥ grade 2;
5. Patients with confirmed HIV infection. HIV testing is not mandatory.
6. Prior history of malignancy except for basal cell carcinoma or carcinoma in situ of the cervix, and with the exception of other malignancies after curative treatment with an interval of at least 3 years.
7. Lactating or pregnant woman, woman of child-bearing potential who do not agree to the usage of highly effective contraception methods (allowed methods of contraception, meaning methods with a rate of failure of less than 1% per year are implants, injectable contraceptives, combined oral contraceptives, intrauterine devices (only hormonal devices), sexual abstinence or vasectomy of the partner). Woman of childbearing potential must have a negative pregnancy test (serum β-HCG) at visit 1.
8. Any other chemotherapy at start;
9. Treatment with other experimental drugs during the course of the study or within the last 30 days or 7 half-lifes, whatever is of longer duration, prior study start;
10. Any psychiatric illness that would affect the patient's ability to understand the demands of the clinical trial;
11. Parallel participation in another clinical trial or participation in another clinical trial within the last 30 days or 7 half-lifes, whatever is of longer duration, prior study start;
12. Patient has already been included in this trial;
13. Patients who do not understand the nature, the scope and the consequences of the clinical trial;
14. Affected persons who might be dependent on the sponsor or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11; Primary Completion 2017-03-28 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
pathologic complete remission rate (pCR rate) | 12 weeks (after 3 cycles and surgery) after enrollment
  The primary objective of the study is to assess the pathologic complete remission rate after induction therapy with gefitinib d -12 to d-1 followed by docetaxel 75 mg/m2 and cisplatin 50 mg/m2 d1+2 q21 and intercalated gefitinib 250 mg d4 to d20 (cycle 1 and 2) and d4-17 (for cycle3), in order to demonstrate feasibility and efficacy of this treatment scheme. It is expected to achieve a pCR ≥30% regression grade IIB and III (Junker criteria) compared to historical controls in the mediastinal lymph nodes.

SECONDARY OUTCOMES:
Adverse Events (AEs) / Serious adverse events (SAEs) | 30 months
  AEs/SAEs from 21 patients during induction CTx with docetaxel and cisplatin in combination with intercalated gefitinib
Surgical R0 resection rate | 30 month
  R0 resection rate as assessed according to the German S3 guidelines
Response: radiologic response based on CT | 30 month
progression free survival (PFS) | 30 month
  Progression-free survival (PFS) will be defined as the time from enrollment to the time of disease progression or relapse or death, or to the date of last assessment without any such event (censored observation).
Overall survival (OS) | 30 month
  The duration of overall survival (OS) will be determined by measuring the time interval from enrollment to the date of death or last observation (censored).
relapse pattern | 30 month
  After the end of treatment will be performed every 3 month (+/- 14 days) for minimum 12 months in order to collect information on relapse and site of relapse
quality of life | 30 month
  Explorative analysis of health related quality of life, QoL at various time points throughout the study, to assess the QoL during and after induction therapy with gefitinib, after three cycles of chemotherapy with intercalated gefitinib including pre- and post surgery
translational research | 30 month
  To collect and store tumor tissue as well as plasma and serum samples for exploratory analyses of potential predictive markers, monitoring of biomarkers during and after treatment
monitoring of epidermal growth factor receptor (EGFR) mutation status | 30 month
  analysis of EGFR ctDNA in patient plasma; screening for EGFR mutation status (activating and resistance mutations especially T790M), monitoring of EGFR mutation status by means of Circulating tumor DNA (ctDNA) detection in patient plasma

CONTACTS AND LOCATIONS:
Overall Officials: Frank Griesinger, Prof. Dr., Principal Investigator — Universitätsklinik für Innere Medizin-Onkologie, Pius-Hospital, Oldenburg
Locations (1):
- Pius-Hospital, Oldenburg, Germany

REFERENCES:
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de